CLINICAL TRIAL: NCT06342713
Title: Phase 1a/1b Randomized Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single- and Multiple-Ascending Doses and Food Effect of BGB-45035 in Healthy Participants and Its Safety and Tolerability in Patients With Autoimmune Dermatological Diseases
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single- and Multiple-Ascending Doses and Food Effect of BGB-45035 in Healthy Participants and in Adults With Autoimmune Dermatological Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-45035-101; CTR20243170 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants; Healthy Subjects; Healthy Volunteers; Autoimmune Diseases; Healthy Adult Participants; Atopic Dermatitis; Prurigo Nodularis
Keywords: Healthy Volunteers; Healthy Subjects; Healthy Participants; BGB-45035; Healthy Adult Participants; IL-33-induced skin inflammation; atopic dermatitis; prurigo nodularis; IRAK4; CDAC
MeSH Terms: conditions — Autoimmune Diseases; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The cohorts in Part A, B, and C will be double-blinded, while Parts D, E, and F will be open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A (Single Ascending Dose) (Experimental): Part A is designed to assess the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic profile of BGB-45035 following single-ascending doses (SAD) in healthy participants.
  Interventions: Drug: BGB-45035; Drug: Placebo
- Part B (Multiple Ascending Dose) (Experimental): Part B is designed to assess safety, tolerability, PK, and pharmacodynamic profile after repeated dosing of BGB-45035 in healthy participants.
  Interventions: Drug: BGB-45035; Drug: Placebo
- Part C (Chinese Substudy) (Experimental): Part C is designed to assess safety, tolerability, PK, and pharmacodynamic profile after repeated dosing of BGB-45035 in healthy Chinese participants.
  Interventions: Drug: BGB-45035; Drug: Placebo
- Part D (Food Effect) (Experimental): Part D is designed to assess the effect of food on BGB-45035 exposure.
  Interventions: Drug: BGB-45035
- Part E (AD Cohort E1) (Experimental): AD Cohort E1 is designed to assess the safety, tolerability, and efficacy of a selected dose of BGB-45035 in participants with moderate to severe AD.
  Interventions: Drug: BGB-45035
- Part E (PN Cohort E2) (Experimental): PN Cohort E2 is designed to assess the safety, tolerability, and efficacy of a targeted dose of BGB-45035 in participants with moderate to severe PN.
  Interventions: Drug: BGB-45035
- Part F (Biomarker Cohort) (Experimental): Part F is designed to assess the pharmacodynamic activity of BGB-45035 in the skin of healthy volunteers.
  Interventions: Drug: BGB-45035

INTERVENTIONS:
Drug: BGB-45035 — Administered orally
Drug: Placebo — Administered orally
  Arms: Part A (Single Ascending Dose); Part B (Multiple Ascending Dose); Part C (Chinese Substudy)

SUMMARY:
This study is the first-in-human (FIH) study of BGB-45035. The study will evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of BGB-45035 with both a single dose and multiple doses administered at different dose levels in healthy participants, followed by a Part E to evaluate the safety and tolerability of BGB-45035 in adults with autoimmune dermatological diseases like atopic dermatitis (AD) and prurigo nodularis (PN). An additional biomarker cohort will be evaluated in Part F.

Study details include:

* The study duration will be up to 24 months.
* The treatment duration will be up to 14 days for Parts A-D, up to 12 weeks for Part E, and up to 3 weeks for Part F.
* Safety follow-up 30 days after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria for Parts A-D and Part F:

1. Female or male participants between the ages of 18 and 55 years inclusive (ages 18 and 45 years for Part C).
2. BMI of 18 to 32 kg/m^2; and a total body weight > 50 kg (110 lbs).
3. Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
4. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
5. Nonsterile male participants must be willing to use a highly effective method of birth control and refrain from sperm donation for the duration of the study and for 90 days after the last dose of study drug.
6. Female participants of childbearing potential can only join Part F and must be willing to use a highly effective method of birth control and refrain from egg donation for the duration of the study and for 90 days after the last dose of study drug. They must also have a negative urine pregnancy test at baseline before first dose of study drug.

Inclusion Criteria for Part E

1. Female or male participants between the ages of 18 to 75 years of age.
2. Female participants of childbearing potential must be willing to use a highly effective method of birth control and refrain from egg donation for the duration of the study and for 90 days after the last dose of study drug. They must also have a negative urine pregnancy test at baseline before first dose of study drug.
3. AD Cohort E1:

   1. Chronic AD diagnosed by the Eichenfield revised criteria of Hannifin and Rajka that has been present for at least 1 year before the Screening Visit.
   2. Prior to baseline assessment, participants with AD must have used only nonmedicated topical emollients twice daily for at least 7 days, without any active ingredients or additives that could impact AD treatment (such as hyaluronic acid, urea, ceramide, or filaggrin degradation products). Participant's response to treatment must have remained inadequate at baseline. Additionally, the participant must be willing and able to adhere to standardized background topical therapy as outlined in the protocol throughout the remainder of the study.
4. PN Cohort E2:

   1. Diagnosed as PN by a dermatologist for at least 3 months before the Screening Visit with prurigo lesions on upper limbs with or without lesions on the trunk or lower limbs.
   2. Minimum of 20 PN lesions in total on either of the following: both legs, both arms, and/or the trunk at the Screening Visit and on Day 1.

General Inclusion Criteria:

1. Must agree to avoid prolonged exposure to the sun and not to use tanning booths, sun lamps, or other ultraviolet light sources during the study.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy or cholecystectomy).
3. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product, whichever is longer.
4. 12-lead ECG demonstrating QTcF > 450 milliseconds.
5. Clinically significant abnormality on chest radiograph performed at screening or within 3 months of screening date.
6. History of tuberculosis or active or latent or inadequately treated infection, positive IGRA tests
7. Herbal supplements (including St. John's Wort) and hormone replacement therapy must be discontinued 14 days prior to the first dose of study medication.
8. Vaccination with live virus, attenuated live virus, or any live viral components within the 6 weeks prior to the first dose of study drug or is to receive these vaccines at any time during treatment or within 8 weeks following completion of study treatment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-05-23 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) in Parts A-E | From the first dose of study drug to 30 days after the last dose; up to approximately 44 days for Parts A-D and up to 16 weeks for Part E
Parts A-D: Number of participants with clinically significant changes from baseline in clinical laboratory values | Baseline and up to approximately 1 month
  Laboratory values include hematology, clinical chemistry, coagulation, and urinalysis
Parts A-D: Number of participants with clinically significant changes from baseline in vital signs | Baseline and up to approximately 1 month
  Vital signs include blood pressure and pulse rate
Parts A-D: Number of participants with clinically significant changes from baseline in cardiac conduction intervals | Baseline and up to approximately 1 month
  As assessed via 12-lead electrocardiogram (ECG)

SECONDARY OUTCOMES:
Parts A & D: Area under the plasma concentration time curve from time zero to last quantifiable time (AUClast) of BGB-45035 | Up to approximately 14 days
Parts A & D: Area under the plasma concentration time curve from time zero to infinite time (AUCinf) of BGB-45035 | Up to approximately 14 days
Parts B & C: Area under the plasma concentration time curve from time zero to end of dosing interval (AUCtau) of BGB-45035 | Up to approximately 14 days
Parts A, B, C & D: Maximum observed plasma concentration (Cmax) of BGB-45035 | Up to approximately 14 days
Parts A, B, C & D: Time to maximum plasma concentration (Tmax) of BGB-45035 | Up to approximately 14 days
Parts B & C: Trough plasma concentration (Ctrough) of BGB-45035 | Up to approximately 14 days
Parts A, B, C & D: Half life (t½) of BGB-45035 | Up to approximately 14 days
Parts A, B, & C: Apparent systemic clearance (CL/F) of BGB-45035 | Up to approximately 14 days
Parts A, B, & C: Apparent volume of distribution (Vz/F) of BGB-45035 | Up to approximately 14 days
Parts B & C: Accumulation Ratios of BGB-45035 | Up to approximately 14 days
Part E (AD Cohort E1): Change from baseline in Eczema Area and Severity Index (EASI) score at all scheduled visits | Baseline and up to 16 weeks
Part E (AD Cohort E1): Change from baseline in Investigator Global Assessment (IGA) scale for Atopic Dermatitis (IGA-AD) score at all scheduled visits | Baseline and up to 16 weeks
Part E (PN Cohort E2): Change from baseline in Investigator Global Assessment (IGA) Stage score at all scheduled visits | Baseline and up to 16 weeks
Part E (PN Cohort E2): Change from baseline in Investigator Global Assessment (IGA) Activity score at all scheduled visits | Baseline and up to 16 weeks
Part E: Change from baseline of Peak Pruritus Numerical Rating Scale (PP-NRS) at all scheduled visits | Baseline and up to 16 weeks
Part E: Change from baseline in Average of Pruritus Numerical Rating Scale (AP-NRS) at all scheduled visits | Baseline and up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (13):
- Australia (2):
  - Innovate Clinical Research, Waitara, New South Wales
  - Cmax Clinical Research, Adelaide, South Australia
- China (8):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Hospital of Qingdao University Branch West Coast, Qingdao, Shandong
  - Chengdu Second Peoples Hospital, Chengdu, Sichuan
- New Zealand (3):
  - Optimal Clinical Trials Ltd, Auckland
  - Pacific Clinical Research Network Auckland, Takapuna
  - Lakeland Clinical Trials Wellington, Upper Hutt

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/